CLINICAL TRIAL: NCT06439550
Title: Adjuvant Treatment With Serplulimab，Trastuzumab and SOX in the of HER-2 Positive Gastric/Gastroesophageal Junction Carcinoma (GC/GEJC)
Brief Title: Adjuvant Treatment With Serplulimab，Trastuzumab and SOX in the HER-2 Positive GC/GEJC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Feng Wang, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLX10IIT123
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2023-11

CONDITIONS: HER2-positive Gastric Cancer
MeSH Terms: interventions — Trastuzumab; Oxaliplatin; Tegafur

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Serplulimab，Trastuzumab and SOX (Experimental): Within 4 weeks after surgery, patients will be enrolled in the study and started on Serplulimab (300mg, q3w) + Trastuzumab (First dose 8mg/kg, maintenance 6mg/kg, q3w) + oxaliplatin (130mg/m2, q3w) + Tegafur (40mg/m2, bid d1-d14, q3w). Among them, oxaliplatin + Teggio can be used for 4-6 cycles according to the patient's tolerance, and Serplulimab + trastuzumab can be continued until 12 months or tumor recurrence or metastasis
  Interventions: Drug: Serplulimab; Drug: Trastuzumab; Drug: Oxaliplatin + Tegafur

INTERVENTIONS:
Drug: Serplulimab — 300mg, q3w
Drug: Trastuzumab — First dose 8mg/kg, maintenance 6mg/kg, q3w
Drug: Oxaliplatin + Tegafur — oxaliplatin (130mg/m2, q3w) + Tegafur (40mg/m2, bid d1-d14, q3w).
  Other Names: SOX

SUMMARY:
This is a prospective, single arm, multicenter phase II study to assess the effectiveness of Serplulimab，Trastuzumab and SOX in the adjuvant treatment of HER-2 Positive Gastric/Gastroesophageal Junction Carcinoma (GC/GEJC)

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastric adenocarcinoma/esophagogastric junction adenocarcinoma, HER-3 + or HER-2 +, with Fish amplification;
2. Subjects must complete R0 resection before enrollment；If they received neoadjuvant therapy, it was required that the neoadjuvant therapy regimen should not contain anti-HER-2 targeted drugs;
3. Postoperative pathology: II-III;
4. Age 18-75 years old;
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
6. Blood routine and biochemistry within 7 days before enrollment : a. Hemoglobin ≥90g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelets ≥100×109/L (no blood transfusion within 14 days before treatment, no granulocyte colony-stimulating factor, no correction with other drugs); b. ALT and AST≤2.5 times the normal upper limit (ULN); ALP≤2.5 times ULN; c. Serum total bilirubin <1.5 ULN (Gilbert syndrome patients with total bilirubin <3 ULN can be enrolled); d. Serum creatinine <1.5 ULN or estimated glomerular filtration rate ≥60ml/min/1.73m2; e. Serum albumin ≥30g/L; f. International Normalized Ratio (INR) or prothrombin time (PT) ≤1.5 times ULN, unless the patient is receiving anticoagulant therapy and the PT value is within the intended treatment range of the anticoagulant; g. Activated partial thromboplastin time (APTT) ≤1.5 times ULN.
7. No serious concomitant diseases that make the survival time less than 5 years;
8. Voluntary and able to adhere to the program during the study;
9. Provide written informed consent form before entering the study, and the subjects has understood that he can withdraw from the study at any time during the study without any loss.

Exclusion Criteria:

1. A history of any other malignancy in the past 5 years (except carcinoma in situ or basal cell carcinoma of the skin or squamous cell carcinoma of the skin)；Patients with small gastric stromal tumors and other tumors may be excluded if the researcher determines that other tumors will not affect the patient's life in the short term；
2. Participated in clinical trials of other drugs within four weeks;
3. Have any active autoimmune disease or a history of autoimmune disease (e.g., but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism; subjects has vitiligo; asthma that has completely relieved in childhood and does not require any intervention in adulthood can be included; asthma that requires medical intervention with bronchodilators cannot be included)
4. Requires systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration to treat a current condition.
5. Any active malignant tumour within 2 years, excluding the specific cancer being studied in this trial and the locally recurrent cancer that has been cured (such as basal cell or squamous cell skin cancer that has been removed, superficial bladder cancer cancer, cervical or breast cancer in situ);
6. Subjects with central nervous system metastasis or a history of central nervous system metastasis. With clinically suspected CNS metastasis, CT or MRI must be performed within 28 days before starting treatment to rule out CNS metastasis；
7. With unstable angina pectoris; Newly diagnosed angina pectoris within 3 months prior to screening or myocardial infarction events occurred within 6 months prior to screening; Arrhythmias (including QTcF: ≥ 450 ms for males and ≥ 470 ms for females) require long-term use of antiarrhythmic drugs and a New York Heart Association grade of ≥ II cardiac dysfunction;
8. Or urinary protein qualitative ≥2+, 24 hours urinary protein > 1g
9. For female subjects: should be surgically sterilized, postmenopausal, or consent to use a medically approved contraceptive during the study treatment period and for 6 months after the end of the study treatment period; Serum or urine pregnancy tests must be negative within 7 days before enrollment and must be non-lactating. Male subjects: patients who should be surgically sterilized or who have consented to use a medically approved contraceptive method during the study treatment period and for 6 months after the end of the study treatment period;
10. Liver transplantation patients；
11. With infectious pneumonia, non-infectious pneumonia, interstitial pneumonia and other subjects require the use of corticosteroids;
12. Have a history of chronic autoimmune diseases, such as systemic lupus erythematosus;
13. Have a history of inflammatory bowel diseases such as ulcerative colitis and Crohn's disease, and a history of chronic diarrhea diseases such as irritable bowel syndrome；
14. Have a history of sarcoidosis or tuberculosis；
15. With active HBV, HCV，and HIV infection；
16. Subjects with a history of psychotropic substance abuse and are unable to abstain or have mental disorders; 17) Thoracic or abdominal effusion with clinical symptoms that require clinical intervention; 18) A history of immunodeficiency, or other acquired or congenital immunodeficiency diseases, or a history of organ transplantation; 19) According to the judgment of the researcher,there is a serious concomitant disease that endangers the patient's safety or interferes with the patient's completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease progression free survival （DFS） | 24 months after the last subject participating in
  Objective response rate according to RECIST 1.1

SECONDARY OUTCOMES:
Overall survival (OS） | 24 months after the last subject participating in
  Overall survival
Recurrence rate | 24 months after the last subject participating in
  Objective response rate according to RECIST 1.1
Safety and tolerability based on incidence of treatment-emergent adverse events as assessed by CTCAE | through study completion, an average of 1 year
  Safety and tolerability based on incidence of treatment-emergent adverse events as assessed by CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — The First Affiliated Hospital of Zhengzhou University

IPD SHARING:
Plan to Share IPD: No